CLINICAL TRIAL: NCT04104139
Title: Phase 1b Study to Assess the Safety of Neoadjuvant TAS-102 (Trifluridine/Tipiracil) With Concurrent Radiation in Previously Untreated Resectable Stage II and Stage III Rectal Cancer (FIERCE)
Brief Title: TAS-102 With Concurrent Radiation for the Treatment of Untreated Resectable Stage II-III Rectal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Charles D Lopez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019576; NCI-2019-06387 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-19069-L; STUDY00019576 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Rectal Adenocarcinoma; Stage IIA Rectal Cancer AJCC v8; Stage IIB Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TAS-102, IMRT, 3D-CRT) (Experimental): Patients receive TAS-102 PO BID Monday-Friday on weeks 1, 3, and 5. Patients also undergo IMRT or 3D-CRT 5 days per week on weeks 1-5. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care FOLFOX or CAPOX.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102

SUMMARY:
This phase 1b trial studies the side effects and best dose of TAS-102 when given together with radiation therapy in treating patients with stage II-III rectal cancer that has not been treated and can be removed by surgery (resectable). Drugs used in chemotherapy, such as TAS-102, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. This study is being done to find out the safest dose of TAS-102 that can be used with radiation treatment for rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase 2 dose of trifluridine and tipiracil hydrochloride (TAS-102) per the proportion of grade 3 or higher adverse events during chemo-radiation therapy (CRT) with concurrent TAS-102 at the maximum tolerated dose by allowing no more than 30% grade 3 or higher adverse events.

SECONDARY OBJECTIVES:

I. Evaluate safety of participants treated with TAS-102 during radiation therapy (RT).

II. Evaluate treatment emergent adverse events (TEAEs) attributable to TAS-102 with RT during fluorouracil/leucovorin calcium/oxaliplatin (FOLFOX) or capecitabine/oxaliplatin (CAPOX) treatment.

EXPLORATORY OBJECTIVES:

I. To preliminary assess the rates of complete clinical response (cCR) by magnetic resonance imaging (MRI) and by endoscopy after TAS-102 with concurrent CRT.

II. To preliminary assess the rates of cCR by MRI and by endoscopy after treatment with FOLFOX.

III. To preliminary assess the rates of pCR after standard total mesorectal excision (TME).

OUTLINE: This is dose-escalation study of TAS-102.

Patients receive TAS-102 orally (PO) twice daily (BID) Monday-Friday on weeks 1, 3, and 5. Patients also undergo intensity modulated radiotherapy (IMRT) or 3-dimensional conformal radiotherapy (3D-CRT) 5 days per week on weeks 1-5. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care FOLFOX or CAPOX.

After completion of study treatment, patients are followed for up to a total of 16 weeks (3 months) from end of FOLFOX or CAPOX treatment until rectal cancer surgery or death, whichever occurs first. Participants that opt for a non-surgical option at the end of chemotherapy may be followed for a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* All races and ethnic groups will be included
* Histologically confirmed diagnosis of adenocarcinoma of the rectum
* Clinical stage II (T3-4aN0M0) and stage III (T1-4aN1+M0) based on MRI
* Resectable primary rectal tumor at baseline
* No evidence of distant metastases
* No prior pelvic radiation therapy
* No prior chemotherapy or surgery for rectal cancer
* No active infections requiring systemic antibiotic treatment (oral antibiotics are acceptable at the discretion of the treating physician)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Hemoglobin >= 9.0 gm/dL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits, OR creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A female of childbearing potential is defined of one who is biologically capable of becoming pregnant. Reliable contraception should be used starting from trial screening and must be continued throughout the study
* Females of childbearing potential must agree to use effective contraceptive method starting with the first dose of study therapy through 6 months after the last dose of study therapy
* Male participants must agree to use an effective method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy
* Participants must read, have the ability to understand, agree to, and sign a statement of Informed Consent prior to participation in this study
* Participants must, as part of their planned treatment per institutional guidelines, be:

  * Scheduled to receive preoperative FOLFOX or CAPOX chemotherapy, which requires a central venous access device for administration
  * Able to undergo planned TME of the rectal tumor per institutional standards

Exclusion Criteria:

* Recurrent rectal cancer
* Primary unresectable rectal cancer. A tumor is considered unresectable when invading adjacent organs (T4b disease) and an en bloc resection will not achieve negative margins. Rectal cancer presenting with concurrent or overlapping sites in the colon is eligible if these sites could be removed with surgery
* Distant nodal disease (retroperitoneal nodes), or any metastatic disease by computed tomography (CT) or positron emission tomography (PET)
* Creatinine > 1.5 x ULN
* History of peripheral neuropathy > grade 2
* History of malabsorption syndromes or inflammatory bowel disease
* Use of immunosuppressive or myelosuppressive medications including but not limited to adalimumab, azathioprine, BCG, clozapine, cyclosporine, deferiprone, etanercept, fingolimod, hydroxyurea, interferon, leflunomide, methotrexate, mycophenolate, natalizumab, pimecrolimus, rituximab, sirolimus, and tacrolimus
* Inability to take oral medications
* Participants who received prior pelvic radiotherapy
* Use of induction chemotherapy prior to chemo-radiation of rectal cancer
* Use of other chemotherapy regimens other than FOLFOX or CAPOX
* Participants who are unable to undergo an MRI
* Participants who are unable to undergo TME
* Refusal of standard-of-care TME of the rectal tumor if there is persistent disease after neoadjuvant treatment
* Participants with a history of any arterial thrombotic event within the past 6 months, including angina (stable or unstable), myocardial infarction (MI), transient ischemic attack (TIA), or cerebrovascular accident (CVA)
* Participants with a recent history of venous thrombotic episodes such as deep venous thrombosis and pulmonary embolism within the past 3 months. If these episodes occurred more than three months prior to enrollment, they may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Similarly, participants who are anticoagulated for atrial fibrillation or other conditions may participate, provided they are on stable doses of anticoagulant therapy
* Febrile illness within 7 days of study enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102 or other agents used in this study
* Other anticancer or experimental therapy. No other experimental therapies including for other disease indications are allowed while the participant is receiving study treatment
* Women who are pregnant or breast-feeding
* Participants with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study
* Participants with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of dose limiting toxicity (DLT)s for TAS-102 at the maximum tolerated dose (MTD) | Up to end of week 8, or start of fluorouracil/leucovorin calcium/oxaliplatin (FOLFOX) or capecitabine/oxaliplatin (CAPOX) chemotherapy, whichever occurs first
  Will be assessed through the Bayesian optimal interval design and will be determined by the proportion of grade 3 or higher adverse events during chemo-radiation therapy (CRT) with TAS-102 at the MTD by allowing no more than 30% DLT. The proportion will be descriptively noted.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) (all grade) for TAS-102 concurrent with radiation therapy (RT) | Up to start of FOLFOX or CAPOX (up to 8 weeks)
  Descriptive statistics of safety will be presented using National cancer Institute Common Terminology Criteria for Adverse Events version 5.0., with AEs tabulated by the MedDRA preferred term and system organ class. The incidence of AEs (all grades) for TAS-102 with concurrent RT will be assessed using the CRT analysis set.
Incidence of grade 3 or higher treatment emergent adverse events (TEAEs) during FOLFOX or CAPOX treatment | Up to end of FOLFOX or CAPOX (up to 16 weeks)
  The incidence of grade 3 or higher TEAEs during FOLFOX or CAPOX chemotherapy will be assessed using the FOLFOX/CAPOX analysis set.

OTHER OUTCOMES:
Rate of complete response (CR) by magnetic resonance imaging (MRI) after chemo-radiation therapy (CRT) | Prior to starting FOLFOX or CAPOX regimen (up to 8 weeks)
  MRI report after CRT will be collected from medical records. Discrepancies will be resolved with the diagnostic radiology investigators of the research team. Complete response based on MRI will be tabulated as proportions and analyzed descriptively using the CRT analysis sets.
Rate of CR by endoscopic exam after CRT | Prior to starting FOLFOX or CAPOX regimen (up to 8 weeks)
  Endoscopic exam report after CRT will be collected from medical records (as available). Discrepancies will be resolved with the surgical oncology investigators of the research team. Complete response based on endoscopic exam will be tabulated as proportions and analyzed descriptively using the CRT analysis sets.
Rate of clinical complete response (cCR) by MRI and endoscopic response after CRT | Prior to starting FOLFOX or CAPOX regimen (up to 8 weeks)
  cCR requires CR for MRI and CR for endoscopic responses. The number of cCR after CRT will be tabulated as proportions using the CRT analysis sets, respectively.
Rate of CR by MRI after CRT and FOLFOX or CAPOX | At end of chemotherapy visit (up to 21 weeks)
  MRI report after CRT + FOLFOX or CAPOX will be collected from medical records. Discrepancies will be resolved with the diagnostic radiology investigators of the research team. Complete response based on MRI will be tabulated as proportions and analyzed descriptively using the CRT and the FOLFOX/CAPOX analysis sets, respectively.
Rate of CR by endoscopic exam after CRT and FOLFOX or CAPOX | At end of chemotherapy visit (up to 21 weeks)
  Endoscopic exam report after CRT + FOLFOX or CAPOX will be collected from medical records (as available). Discrepancies will be resolved with the surgical oncology investigators of the research team. Complete response based on endoscopic exam will be tabulated as proportions and analyzed descriptively using the CRT and the FOLFOX/CAPOX analysis sets, respectively.
Rate of cCR by MRI and endoscopic response after CRT and FOLFOX or CAPOX | At end of chemotherapy visit (up to 21 weeks)
  cCR requires CR for MRI and CR for endoscopic responses. The number of cCR after CRT and after CRT + FOLFOX or CAPOX will be tabulated as proportions using the CRT and the FOLFOX/CAPOX analysis sets, respectively.
Rate of pathologic complete response after standard total mesorectal excision (TME) | At resection (up to 29 weeks)
  Pathology report after standard TME will be collected from medical records. Discrepancies will be resolved with the surgical oncology and pathology investigators of the research team. Complete response based on pathology will be tabulated as proportions and analyzed descriptively using the TME population.

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Lopez, MD, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States